CLINICAL TRIAL: NCT01385904
Title: Plasma Concentrations of Ketamine and Norketamine in Patients Using Topical Application of 10% Ketamine for Neuropathic Pain.
Brief Title: Blood Levels of Ketamine in Patients Using Topical Application of 10% Ketamine Gel for Neuropathic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Dr. Patricia Morley-Forster, University of Western Ontario
Other Study IDs: R-11-137; 17756 (Other: REB)
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Neuropathic Pain.
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to measure how much, if any, ketamine is absorbed into the blood stream after ketamine gel is applied to the skin. The investigators expect that the topical administration will provide pain relief locally, at the site of pain, but not be absorbed into the bloodstream and thus not cause side effects. This research will help assess the safety of this drug by measuring the blood concentrations of the drug.

Ketamine is a general anesthetic drug but also has excellent pain relieving qualities. It has been used to relieve chronic pain by administering intravenously, by mouth, or as an injection beneath the skin. When given these ways ketamine can occasionally cause side effects like dizziness, nausea, nightmares, agitation, hallucinations. Recently it has been used topically for patients with neuropathic pain in order to avoid the dizziness and nausea side effects.

Neuropathic Pain can be partially caused by the misfiring of small nerve fibers close to the area of pain. By applying it on the skin, it is expected the drug can penetrate the skin and act directly on the small nerve fibers. The advantage is that less drug will get into the blood circulation. Up to now, it has not been carefully studied how much of the drug appears in the circulation after application on the skin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral, focal neuropathic pain such as or complex regional pain syndrome following surgery, bony, soft tissue trauma or nerve trauma, associated with significant allodynia and hyperalgesia who score equal to or greater than 4 in the DN4 questionnaire.
* Duration of pain more than 3 months.
* Ability to speak English adequately to consent to and participate in the study

Exclusion Criteria:

* Allergy to ketamine
* Severe medical illnesses like, e.g. unstable angina, tachyarryhthmias, renal or hepatic failure
* History of psychosis.
* Patients who are already on oral ketamine treatment.
* Patients who are taking HIV Antiretrovirals: (indinavir, nelfinavir, ritonavir saquinavir); Antibiotics: (clairithromycin, itraconazole, ketoconazole, telithromycin,fluconazole, erythromycin); Calcium Channel Blockers (verapamil, diltiazem),Amiodarone, Ciprofloxacin. (These drugs inhibit CYP 3A4 enzyme which metabolises ketamine)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the St Josephs Hospital pain clinic with chronic neuropathic pain.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Morley- Forster, MD, FRCPC, Principal Investigator — Western University, Canada
Locations (1):
- Pain Clinic, St. Joseph's Health Care London Hospitals, London, Ontario, Canada

REFERENCES:
- [Background] Poyhia R, Vainio A. Topically administered ketamine reduces capsaicin-evoked mechanical hyperalgesia. Clin J Pain. 2006 Jan;22(1):32-6. doi: 10.1097/01.ajp.0000149800.39240.95. PMID 16340591
- [Background] Finch PM, Knudsen L, Drummond PD. Reduction of allodynia in patients with complex regional pain syndrome: A double-blind placebo-controlled trial of topical ketamine. Pain. 2009 Nov;146(1-2):18-25. doi: 10.1016/j.pain.2009.05.017. Epub 2009 Aug 22. PMID 19703730
- [Background] Zapantis G, Csoka I, Csanyi E, Horvath G, Eros I. Evaluation of ketamine systemic absorption from topical preparations. Short Communication. Acta Biol Hung. 2006 Sep;57(3):387-9. doi: 10.1556/ABiol.57.2006.3.12. PMID 17048702
- [Background] Clements JA, Nimmo WS, Grant IS. Bioavailability, pharmacokinetics, and analgesic activity of ketamine in humans. J Pharm Sci. 1982 May;71(5):539-42. doi: 10.1002/jps.2600710516. PMID 7097501
- [Background] Pedersen JL, Galle TS, Kehlet H. Peripheral analgesic effects of ketamine in acute inflammatory pain. Anesthesiology. 1998 Jul;89(1):58-66. doi: 10.1097/00000542-199807000-00011. PMID 9667294
- [Background] Lynch ME, Clark AJ, Sawynok J, Sullivan MJ. Topical 2% amitriptyline and 1% ketamine in neuropathic pain syndromes: a randomized, double-blind, placebo-controlled trial. Anesthesiology. 2005 Jul;103(1):140-6. doi: 10.1097/00000542-200507000-00021. PMID 15983466
- [Background] Grant IS, Nimmo WS, Clements JA. Pharmacokinetics and analgesic effects of i.m. and oral ketamine. Br J Anaesth. 1981 Aug;53(8):805-10. doi: 10.1093/bja/53.8.805. PMID 7272143